CLINICAL TRIAL: NCT06682806
Title: A Phase 2, Safety and Efficacy Study of PRT3789 in Combination With Pembrolizumab in Patients With Advanced or Metastatic Solid Tumors With a SMARCA4 Mutation
Brief Title: A Study of PRT3789 in Combination With Pembrolizumab in Patients With Advanced or Metastatic Solid Tumors With a SMARCA4 Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Prelude Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT3789-02; KEYNOTE-G02 (Other: Merck Sharp and Dohme LLC); MK-3475-G02 (Other: Merck Sharp and Dohme LLC); 2024-516889-11-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-29; First posted 2024-11-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Esophageal Cancer; Metastatic Solid Tumor; Non-small Cell Lung Cancers; SMARCA4 Gene Mutation
Keywords: Advanced Solid Tumors; BRG1; BRM; Esophageal Cancer; Metastatic Solid Tumors; Non-Small Cell Lung Cancers; NSCLC; PRT3789; Pembrolizumab; Keytruda®; SMARCA2 Degrader; SMARCA4
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT3789/Pembrolizumab combination (Experimental): PRT3789 is administered as an intravenous infusion once weekly for 3 weeks; Pembrolizumab is administered at 200 mg as an intravenous infusion over 30 min every 3 weeks
  Interventions: Drug: PRT3789; Drug: pembrolizumab

INTERVENTIONS:
Drug: PRT3789 — PRT3789 is administered as an intravenous infusion once weekly for 3 weeks
Drug: pembrolizumab — Pembrolizumab is administered at 200 mg as an intravenous infusion over 30 min every 3 weeks
  Other Names: KEYTRUDA®

SUMMARY:
This is a Phase 2 an open-label, multi-center study to determine the safety, tolerability, efficacy, pharmacokinetics, pharmacodynamics, and anti-tumor activity of PRT3789 in combination with pembrolizumab in patients with advanced, recurrent or metastatic solid tumors with a SMARCA4 mutation.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase 2 study of PRT 3789, a first-in-class SMARCA2 targeted protein degrader, in combination with pembrolizumab, a potent humanized immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD-1) receptor, evaluating patients with Advanced or Metastatic Solid Tumors with a SMARCA4 Mutation. This study consists of 2 parts. Part 1 is a safety run-in and will establish the dose of PRT3789 to be used in combination with pembrolizumab in the main study (Part 2). For Part 2 (Main study) primary endpoints are ORR (defined as the proportion of patients with a confirmed best overall response of either complete response or partial response) and duration of response per investigator assessment per RECIST v1.1.

Approximately 46 to 60 patients will be enrolled in Part 1 and Part 2 based on the dose of PRT3789 selected/cleared during the safety run-in.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures, including providing informed consent.
* Patients must either progress on standard of care therapy or be ineligible for standard of care therapy in order to be eligible for enrollment on the study.
* Part 1 Safety Run-in: Patients with advanced, recurrent, or metastatic histologically or cytologically confirmed solid tumor malignancy and any mutation of SMARCA4 detected by next generation sequencing in tumor tissue or blood, or absence of SMARCA4 protein (BRG1). Part 2 Main Study: Patients with advanced, recurrent, or metastatic histologically confirmed esophageal cancer or NSCLC and have a deleterious SMARCA4 mutation, or absence of SMARCA4 protein (BRG1) detected by immunohistochemistry in tumor tissue using a clinically validated laboratory test.
* Part 1 Run-in: Measurable or non-measurable (but evaluable) disease per RECIST v1.1 as assessed by the local site investigator/radiologist. Part 2 Main Study: Measurable disease per RECIST v1.1 as assessed by the local site investigator/radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.
* Willingness and ability to provide tumor tissue (i.e., archived or fresh tumor biopsy if archived tumor tissue is unavailable)
* Adequately controlled blood pressure with or without antihypertensive medications.
* Patients with HIV must have well-controlled HIV on antiretroviral therapy.
* Adequate organ function

Exclusion Criteria:

* Patients who have adverse events due to previous anticancer therapies and/or complications from prior surgical intervention must have recovered to ≤ Grade 1 or baseline before starting study treatment. Patients with endocrine-related AEs who are adequately treated with hormone replacement or patients who have ≤ Grade 2 neuropathy are eligible.
* Other acute or chronic medical or psychiatric conditions that would make the patient inappropriate for entry into this study.
* Patients with solid tumors with a known concomitant SMARCA2 mutation or loss of protein expression.
* Uncontrolled or symptomatic central nervous system (CNS) metastases or leptomeningeal disease and/or carcinomatous meningitis).
* History of or current (noninfectious) pneumonitis/interstitial lung disease
* Diagnosis of immunodeficiency disease/disorder.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Patients who received prior treatment with an agent directed to a stimulatory or co-inhibitory T-cell receptor.
* Currently taking a strong or moderate CYP3A4 inhibitor or inducer and St. John's Wort and are unable to discontinue use within 15 days of the first dose of study treatment.
* Receipt of any targeted therapy directed against BRM/BRG1 (SMARCA2/SMARCA4).
* Pregnant or breastfeeding or plan to become pregnant during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PRT3789 in combination with pembrolizumab as measured by incidence of DLTs (Part 1) | Baseline through completion of study, an average of 2 years
  Safety and tolerability will be evaluated by incidence of dose-limiting toxicities (DLTs)
Safety and tolerability of PRT3789 in combination with pembrolizumab as measured by incidence and severity of AEs according to NCI CTCAE (Part 1) | Baseline through study completion, an average of 2 years
  Safety and tolerability will be evaluated by incidence and severity of adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Efficacy of PRT3789 in combination with pembrolizumab in patients with advanced or metastatic esophageal or NSCLC and deleterious SMARCA4 mutation: Objective Response Rate (Part 2) | Baseline through study completion, an average of 2 years
  Objective response rate defined as the proportion of patients with a confirmed best overall response of either complete response or partial response, as determined per investigator assessment by RECIST v1.1
Efficacy of PRT3789 in combination with pembrolizumab in patients with advanced or metastatic esophageal or NSCLC and deleterious SMARCA4 mutation: Duration of Response (Part 2) | Baseline through study completion, an average of 2 years
  Duration of response defined as the time from the date of the first documented response (complete response or partial response) to the earliest date of disease progression, as determined per investigator assessment by RECIST v1.1, or death due to any cause

SECONDARY OUTCOMES:
Efficacy of PRT3789 in combination with pembrolizumab: Objective Response Rate (Part 1) | Baseline through study completion, an average of 2 years
  Objective response rate defined as the proportion of patients with a confirmed best overall response of either complete response or partial response, as determined per investigator assessment by RECIST v1.1
Efficacy of PRT3789 in combination with pembrolizumab: Duration of Response (Part 1) | Baseline through study completion, an average of 2 years
  Duration of response defined as the time from the date of the first documented response (complete response or partial response) to the earliest date of disease progression, as determined per investigator assessment by RECIST v1.1, or death due to any cause
Efficacy of PRT3789 in combination with pembrolizumab (part 1 and part 2): Clinical Benefit Response | Baseline through study completion, an average of 2 years
  Clinical benefit response defined as the proportion of patients with a best overall response of complete response, partial response, or durable stable disease (24 weeks or longer), as determined per investigator assessment by RECIST v1.1
Efficacy of PRT3789 in combination with pembrolizumab (part 1 and part 2): Progression-Free Survival | Baseline through study completion, an average of 2 years
  PFS defined as the time from the date of first dose of investigational product to the date of first documented progressive disease, as determined per investigator assessment by RECIST v1.1, or death due to any cause
Efficacy of PRT3789 in combination with pembrolizumab (part 1 and part 2): Overall Survival | Baseline through study completion, an average of 2 years
  Overall survival defined as the time from the date of first dose of investigational product to death due to any cause
Safety and tolerability of PRT3789 in combination with pembrolizumab as measured by AEs according to NCI CTCAE | Baseline through study completion, an average of 2 years
  Safety and tolerability will be evaluated by incidence and severity of adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Safety and tolerability of PRT3789 in combination with pembrolizumab: as measured by key clinical laboratory parameters | Baseline through study completion, an average of 2 years
  Laboratory shift tables reflecting mean and CTCAE grade changes from baseline values for key laboratory analytes of alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, creatinine, hemoglobin, platelet count, neutrophil count, lymphocyte count, and leukocyte count
Safety and tolerability as measured by incidence of dose modification due to AEs | Baseline through study completion, an average of 2 years
  Safety and tolerability will be evaluated by dose interruption, modification, and discontinuation due to adverse events (AEs)
PK profile of PRT3789 in combination with pembrolizumab: Maximum observed plasma concentration: Maximum observed plasma concentration | Baseline through study completion, an average of 2 years
  Pharmacokinetics will be calculated including the maximum observed plasma concentration
PK profile of PRT3789 in combination with pembrolizumab: Area under the curve | Baseline through study completion, an average of 2 years
  Pharmacokinetics will be calculated including the area under the plasma concentration versus time curve (AUC)
PK profile of PRT3789 in combination with pembrolizumab: Time of maximum concentration (Tmax) and half-life (T1/2) | Baseline through study completion, an average of 2 years
  Pharmacokinetic parameters will be calculated using standard non-compartmental techniques

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, PLLC - Greco-Hainsworth Centers for Research, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (3):
  - IOB - Next Oncology - Hospital Quironsalud Barcelona, Barcelona
  - START Barcelona - HM Nou Delfos, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz - Servicio de Oncologia, Madrid